CLINICAL TRIAL: NCT03087045
Title: Behavioral Manifestations of Listening Effort
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hillary A Snapp, Assistant Professor, University of Miami
Other Study IDs: 20170031
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Listening Effort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this investigation is to investigate the behavioral manifestations of listening effort. Quantifying listening effort based on an easy to measure behavioral metric would allow for better understanding of the effort that goes into processing conversational speech. The investigators hypothesize that the behavior modifications required to improve the signal to noise ratio in increasingly complex listening environments significantly deviates from quiet listening environments. Further, the investigators hypothesize that this directly contributes to increased listening effort and reduced ability to accurately monitor content for everyday conversation.

DETAILED DESCRIPTION:
Listening Effort has been described as a reflection of the cognitive resources necessary for speech understanding. Measures can broadly be classified into Subjective, Physiological and Behavioral measures of Listening Effort (LE). Subjective measures of LE involve the listener rating or answering a questionnaire on the presented auditory stimuli. Some examples of Subjective measures are the multidimensional speech, spatial and qualities (SSQ) scale and Listening effort rating scale. However, these measures suffer from individual bias, for example, what one person might find takes more effort, another might not.

Physiological measures establish relationships between changes in the central and/or autonomic nervous system activity and LE. Effect of LE on central nervous system activity include methods such as using Functional Magnetic Resonance Imaging (fMRI) to compare processing of noise vocoded versus clear sentence stimuli and using Electroencephalography (EEG) to monitor memory/cognitive load. Some methods of measuring effects on Autonomic Nervous system are through Pupillometry and Skin Conductance. Research has found that fluctuating pupil size may be an indicator of mental task load and/or attention, stress and memory. Furthermore, Pupillometric methods have been used to correlate changing measures like pupil size and listening tasks. There are some drawbacks of using pupillometry to measure LE- Absolute pupil size and change in pupil size for presented speech change according to the age of the listener. For instance, Older adults have been found to have smaller absolute pupil size and show lesser change in pupil size when moving from difficult to easier listening conditions. These drawbacks can be accounted for by normalizing the pupil size.

Behavioral measures take into account that the there is a decline in cognitive functions over prolonged mental effort used an auditory dual task paradigm where the primary task was word recognition and the secondary tasks were memory recall and Visual Response times. Apart from the Dual tasks, participants were also asked to assign a subjective rating based on SSQ. Findings revealed 1) that there is empirical evidence linking repeated instances of effortful listening and subsequent cognitive failure and 2) self- report measures did not show the same changes as the behavioral measures. It has been suggested that this may indicate that subjective (self-report) measures and behavioral measures assess separate aspects of fatigue. It may also be due to subjective measures having individual biases.

As mentioned above, there are numerous studies of subjective, objective and behavioral measures of LE, yet, there are no studies of the actual behavior employed by listeners to reduce listening effort. Further, researchers do not understand how these behaviors influence the ability of the listener to monitor and maintain conversational speech. Listeners must rely on both peripheral and central auditory mechanisms to process speech. As the auditory signal increases in complexity, likewise there is an increase in the auditory processing required to understand speech. The effort that the auditory system must put forth to process complex signals is even greater if the signal degraded or imbedded in competing signals such as background noise. This requires increased exertion and mental effort on the part of the listener, and results in a reduction in ability to maintain focus and an increase in fatigue. These issues are further amplified in the presence of a peripheral hearing disorder as listeners do not have the mechanisms required to properly process even simple and unchallenged auditory signals. Research has demonstrated decreasing word recognition accuracy with decreasing Signal to Noise Ratio (SNR) and demonstrated an increase in listening effort when speech was presented in increasingly negative SNRs. Numerous studies have reported on the increase in listening effort required for individuals with hearing loss.

The purpose of this investigation is quantify listening effort based subjective, objective and behavioral measures at different Signal to Noise Ratios (SNR).

ELIGIBILITY:
Inclusion Criteria:

* Normal Hearing

Exclusion Criteria:

* Do not meet inclusion criteria
* Pregnant women
* Prisoners
* Does not speak English
* Those displaying cognitive impairment (Potential study subjects will be screened for potential cognitive impairments that may negatively influence control data. We will use the validated mini mental exam)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be selected from the University of Miami Ear Institute
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-03-18 (Actual); Study Completion 2017-03-18 (Actual)

PRIMARY OUTCOMES:
Evaluate behavior modifications employed by listeners to optimize the signal to noise ratio and decrease listening effort in complex listening environments. | One hour
  We will evaluate compensatory strategies required by listeners to optimize listening in negative signal to noise ratios
Identify correlations in Listening effort measured using Pupillometry | One hour
  Pupillometry has been shown to be an accurate objective measure of listening effort. We will compare the behavioral responses of increased listening effort to physiologic response as measured by change in pupil size

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Snapp, AuD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Department of Otolaryngology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Downs DW. Effects of hearing and use on speech discrimination and listening effort. J Speech Hear Disord. 1982 May;47(2):189-93. doi: 10.1044/jshd.4702.189. PMID 7176597
- [Background] Noble W, Gatehouse S. Effects of bilateral versus unilateral hearing aid fitting on abilities measured by the Speech, Spatial, and Qualities of Hearing Scale (SSQ). Int J Audiol. 2006 Mar;45(3):172-81. doi: 10.1080/14992020500376933. PMID 16579492
- [Background] Hick CB, Tharpe AM. Listening effort and fatigue in school-age children with and without hearing loss. J Speech Lang Hear Res. 2002 Jun;45(3):573-84. doi: 10.1044/1092-4388(2002/046). PMID 12069009
- [Background] Hornsby BW. The effects of hearing aid use on listening effort and mental fatigue associated with sustained speech processing demands. Ear Hear. 2013 Sep;34(5):523-34. doi: 10.1097/AUD.0b013e31828003d8. PMID 23426091
- [Background] Howard CS, Munro KJ, Plack CJ. Listening effort at signal-to-noise ratios that are typical of the school classroom. Int J Audiol. 2010 Dec;49(12):928-32. doi: 10.3109/14992027.2010.520036. Epub 2010 Nov 4. PMID 21047295
- [Background] Kahneman D. 1973. Attention and Effort, New Jersey: Prentice-Hall Inc.
- [Background] Killion MC, Niquette PA, Gudmundsen GI, Revit LJ, Banerjee S. Development of a quick speech-in-noise test for measuring signal-to-noise ratio loss in normal-hearing and hearing-impaired listeners. J Acoust Soc Am. 2004 Oct;116(4 Pt 1):2395-405. doi: 10.1121/1.1784440. PMID 15532670
- [Background] Koelewijn T, Zekveld AA, Festen JM, Kramer SE. Pupil dilation uncovers extra listening effort in the presence of a single-talker masker. Ear Hear. 2012 Mar-Apr;33(2):291-300. doi: 10.1097/AUD.0b013e3182310019. PMID 21921797
- [Background] Kramer S.E., Lorens A., Coninx F., Zekveld A.A., Piotrowska A. et al. Processing load during listening: The influence of task characteristics on the pupil response. Lang Cognitive Proc, 2012. 28: p.426 - 442.
- [Background] Kuchinsky SE, Ahlstrom JB, Vaden KI Jr, Cute SL, Humes LE, Dubno JR, Eckert MA. Pupil size varies with word listening and response selection difficulty in older adults with hearing loss. Psychophysiology. 2013 Jan;50(1):23-34. doi: 10.1111/j.1469-8986.2012.01477.x. Epub 2012 Nov 15. PMID 23157603
- [Background] Laeng B, Sirois S, Gredeback G. Pupillometry: A Window to the Preconscious? Perspect Psychol Sci. 2012 Jan;7(1):18-27. doi: 10.1177/1745691611427305. Epub 2012 Jan 5. PMID 26168419
- [Background] McGarrigle R, Munro KJ, Dawes P, Stewart AJ, Moore DR, Barry JG, Amitay S. Listening effort and fatigue: what exactly are we measuring? A British Society of Audiology Cognition in Hearing Special Interest Group 'white paper'. Int J Audiol. 2014 Jul;53(7):433-40. doi: 10.3109/14992027.2014.890296. Epub 2014 Mar 27. PMID 24673660
- [Background] Picou EM, Ricketts TA, Hornsby BW. Visual cues and listening effort: individual variability. J Speech Lang Hear Res. 2011 Oct;54(5):1416-30. doi: 10.1044/1092-4388(2011/10-0154). Epub 2011 Apr 15. PMID 21498576
- [Background] Piquado T, Isaacowitz D, Wingfield A. Pupillometry as a measure of cognitive effort in younger and older adults. Psychophysiology. 2010 May 1;47(3):560-9. doi: 10.1111/j.1469-8986.2009.00947.x. Epub 2010 Jan 11. PMID 20070575
- [Background] Wild CJ, Yusuf A, Wilson DE, Peelle JE, Davis MH, Johnsrude IS. Effortful listening: the processing of degraded speech depends critically on attention. J Neurosci. 2012 Oct 3;32(40):14010-21. doi: 10.1523/JNEUROSCI.1528-12.2012. PMID 23035108
- [Background] Zekveld AA, Kramer SE, Festen JM. Pupil response as an indication of effortful listening: the influence of sentence intelligibility. Ear Hear. 2010 Aug;31(4):480-90. doi: 10.1097/AUD.0b013e3181d4f251. PMID 20588118
- [Background] Zekveld AA, Kramer SE, Festen JM. Cognitive load during speech perception in noise: the influence of age, hearing loss, and cognition on the pupil response. Ear Hear. 2011 Jul-Aug;32(4):498-510. doi: 10.1097/AUD.0b013e31820512bb. PMID 21233711